CLINICAL TRIAL: NCT06552260
Title: A Surgical Window of Opportunity Clinical Trial of Troriluzole in Recurrent IDH Wild-Type Glioblastoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ugonma Chukwueke (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Biohaven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ugonma Chukwueke, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-339
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma; Recurrent Glioblastoma; Brain Tumor
Keywords: Glioblastoma; Recurrent Glioblastoma; Brain Tumor; Isocitrate dehydrogenase wild-type Glioblastoma
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Presurgical Troriluzole (Experimental): 18 participants will be randomly assigned to this group and with complete:
  * Baseline visit with assessments and MRI.
  * Cycle 0:
    * Day -6 through Day 0: Predetermined dose of Troriluzole 2x daily.
    * Day 0: pre-op MRI
    * Day 0: standard of care surgical resection of tumor
    * Day 0: post-op MRI
  * Cycle 1 through Cycle 3:
    --Days 1 through 28 of 28 day cycle: Predetermined dose of Troriluzole 2x daily.
  * Cycle 3 through End of Treatment:
    --Days 1 through 28 of 28 day cycle: Predetermined dose of Troriluzole 2x daily.
  * MRIs every 8 weeks while on treatment.
  * End of study visit with MRI
  * Follow up every 3 months for 1 year, and then every 6 months for the next 3 years.
  Interventions: Drug: Troriluzole
- Group B: Surgery + Troriluzole (Experimental): 9 participants will be randomly assigned to this group and with complete:
  * Baseline visit with assessments and MRI
  * Day 0: pre-op MRI
  * Day 0: standard of care surgical resection of tumor
  * Day 0: post-op MRI
  * Cycle 1 through Cycle 3:
    --Days 1 through 28 of 28 day cycle: Predetermined dose of Troriluzole 2x daily.
  * Cycle 3 through End of Treatment:
    --Days 1 through 28 of 28 day cycle: Predetermined dose of Troriluzole 2x daily.
  * MRIs every 8 weeks while on treatment.
  * End of study visit with MRI
  * Follow up every 3 months for 1 year, and then every 6 months for the next 3 years.
  Interventions: Drug: Troriluzole

INTERVENTIONS:
Drug: Troriluzole — Tripeptide prodrug of Riluzole, 100 mg capsule, taken orally per protocol.
  Other Names: Trigriluzole; BHV-4157; FC-4157; 2-Amino-N-({methyl-[(6-trifluoromethoxy-benzothiazol-2-ylcarbamoyl)-methyl]-carbamoyl}-methyl)-acetamide monohydrate monohydrochloride; C15H16F3N5O4S.HCl.H2O

SUMMARY:
This research study is studying troriluzole as a possible treatment for recurrent glioblastoma.

The name of the study drug involved in this research study is:

-Troriluzole (a tripeptide prodrug of riluzole)

DETAILED DESCRIPTION:
This is an open-label, randomized window-of-opportunity study of Troriluzole in participants with surgically accessible, recurrent isocitrate dehydrogenase wild-type (IDH WT) glioblastoma (GBM). Surgical window-of-opportunity clinical trials test how active the investigational drug is on tumors. "Investigational" means that the drug is being studied.

Participants will be randomized using a 2:1 ratio into one of two study treatment groups: Group A versus Group B. Randomization means a participant is placed into a study group by chance. Group A will receive Troriluzole prior to and after standard-of-care tumor resection surgery, while Group B will not receive Troriluzole prior to standard-of-care tumor resection surgery but will receive Troluzole after surgery.

The research study procedures include screening for eligibility, study treatment visits, blood tests, tumor biopsies, Magnetic Resonance Imaging (MRI) scans, and electrocardiograms (ECGs).

It is expected that about 27 participants will take part in this research study

Biohaven Pharmaceuticals is funding this research study by providing study drug.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histopathologically confirmed IDH-wildtype glioblastoma, WHO Grade 4, and variants including gliosarcoma as per WHO 2021 criteria (38).
* Prior treatment with radiotherapy with or without chemotherapy.
* Recurrent or progressive disease with no more than 2 prior relapses.
* Confirmed measurable disease per RANO 2.0 for GBM.
* Tumor is documented as IDH1/2 wildtype by direct DNA sequencing, provided that it is performed in a CLIA/CAP-certified laboratory.
* Availability of archival formalin fixed paraffin-embedded (FFPE) tumor tissue block or 20 unstained FFPE slides (5 μm thick) from any prior surgery for mutation testing and additional sequencing.
* Karnofsky Performance Status of ≥ 60.
* Candidate for surgical resection.
* Tumor tissue extending to cortical gray matter based on MRI.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Women of child-bearing potential (WOCBP), defined as any individual assigned female at birth physiologically capable of becoming pregnant, must use highly effective contraception during study treatment and for 1 month after study discontinuation. Highly effective contraception is defined as either:

  * True Abstinence: When this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception.
  * Sterilization: Surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
  * Male Partner Sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female subjects on the study, the vasectomised male partner should be the sole partner for that participant.
  * A barrier method defined as condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository along with a second contraceptive method as described below:

    * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * Appropriate hormonal contraceptives (including any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent - including oral, subcutaneous, intrauterine
* Male subjects should agree to use a highly effective method of contraception starting with the first dose of study therapy through 3 months after the last dose of therapy. Male subjects must not donate semen for 3 months after the last dose of study treatment.
* Ability to understand and the willingness to sign a written informed consent document. (Providing consents in as many languages as possible is encouraged)

Exclusion Criteria:

* Laboratory values at the Screening Visit:

  * ANC count < 1,500/mm3; growth-factor support within 7 days for filgrastim or other short acting biosimilars or 21 days for pegfilgrastim or other long acting biosimilars to increase the ANC is not allowed.
  * Platelets <100,000/mm3;
  * Hemoglobin < 9 g/dL;
  * Total bilirubin > 2 × the upper limit of normal (ULN) (unless subject has documented history of Gilbert's Syndrome in which case subject may be enrolled if total bilirubin is less than 5 mg/dL, assuming all other criteria are fulfilled);
  * Aspartate aminotransferase (AST [SGOT]) > 1.5 x ULN;
  * Alanine aminotransferase (ALT [SGPT]) > 1.5 x ULN;
  * Serum creatinine > 1.5 mg/dL or a calculated creatinine clearance < 60 mL/min; and
  * Positive serum β-hCG test in any individual assigned female at birth and is of childbearing potential (defined as ≤ 50 years of age, or > 50 years of age with a history of amenorrhea for ≤12 months prior to study entry).
* Has presence of diffuse leptomeningeal disease or extracranial disease.
* Prior treatment with troriluzole or riluzole
* From study treatment initiation, treatment with temozolomide less than 23 days, treatment with CCNU or BCNU less than 42 days, treatment with anti-VEGF therapy such as bevacizumab less than 6 months, or treatment with any cancer-directed systemic therapy less than 4 weeks or 5 half-lives, whichever is shorter. No wash-out period is required from tumor treating fields (TTF).
* Use of any investigational agents within 28 days of baseline or 5 half-lives from study initiation, whichever is shorter.
* Radiotherapy within 12 weeks prior to registration unless new enhancement is outside the radiation field (beyond the high-dose region of 80% isodense line) or evidence of viable tumor on histopathologic sampling.
* Presence of a clinically significant allergy, hypersensitivity, or toxicity of prior therapy, with the exception of alopecia or lymphopenia, that has not resolved to ≤ Grade 1 or pre-treatment baseline, as determined by National Cancer Institute CTCAE v 5.0.
* Major surgery within 28 days prior to initiation of study drug.
* Active or clinically unstable bacterial, viral, or fungal infection requiring systemic therapy.
* Any contraindication to MRI examination.
* Requires medications that are known to be strong inhibitors or inducers of CYP1A2 enzymes or anti-glutamergic agents (e.g., perampanel) or hepatotoxic drugs which may increase the risk of hepatotoxicity (e.g., allopurinol, methyldopa, sulfasalazine). A washout of 10 days or 5 half-lives, whichever is shorter, is required prior to study treatment initiation. Oral contraceptives which contain ethinyl estradiol (moderate CYP1A2 inhibitor) are allowed.
* Pregnant or lactating female.
* History of interstitial lung disease.
* Known history of hepatitis B, human immunodeficiency virus (HIV), or active hepatitis C infection requiring treatment with antiviral therapy. NOTE: HIV testing is not required in the absence of clinical suspicion.
* Any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with the interpretation of study results and, in the Investigator's opinion, would make the subject inappropriate for entry into this study.
* Difficulty swallowing or malabsorption syndrome; refractory nausea and vomiting, chronic gastrointestinal (GI) disease or previous significant bowel resection with clinically significant sequelae that would preclude adequate absorption of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
The effect of troriluzole on high-gamma band power (a measure of neuronal activity) via electrocorticography during surgical resection | At time of surgery
  Data will be summarized using descriptive statistics to compare between participants who received presurgical troriluzole and who did not

SECONDARY OUTCOMES:
Concentrations of Extracellular Glutamate in Resected Tissue by MALDI-MSI | From tumor tissue resected at surgery
  Data will be summarized using descriptive statistics to compare between participants who received presurgical troriluzole and who did not. For MALDI-MSI, raw mass spectrometry data will be analyzed by a combination of Protein Discoverer (Thermo) and in-house software (Computer Assisted Manual Validation, CAMV) to provide accurate identification and quantification of protein phosphorylation sites for each participant sample.
Grade 3-5 Treatment Related Adverse Event | From tumor tissue resected at surgery
  The percentage of participants who experienced a maximum grade 3-5 treatment-related adverse event based on the Common Toxicity Criteria for Adverse events Version 5.0 (CTCAEv5) as reported on case report forms.
Proliferation Rate (Ki-67) in Resected Tissue | From tumor tissue resected at surgery
  Western blot analysis for proliferation (Ki-67) will be summarized using descriptive statistics
Protein Levels of NLGN3 in Resected Tissue | From tumor tissue resected at surgery
  Western blot analysis for NLGN3 will be summarized using descriptive statistics
Protein Levels of Phosphorylated AMPA Receptor Subunits (e.g. GluA2) in Resected Tissue | From tumor tissue resected at surgery
  Western blot analysis for phosphorylated GluA2 will be summarized using descriptive statistics.
Tumor Tissue Concentration of Troriluzole by MALDI-MSI | From tumor tissue resected at surgery
  MALD-MSI analysis for concentration of troriluzole in resected tumor tissue of participants who received presurgical troriluzole

CONTACTS AND LOCATIONS:
Overall Officials: Ugonma Chukwueke, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu
URL: https://www.dfhcc.harvard.edu/research/clinical-research-support/office-of-data-quality/services-support/clinicaltrialsgov-and-ctrp